CLINICAL TRIAL: NCT05320458
Title: Pulmonary Rehabılıtatıon After Chemotherapy In Patıents Wıth Non-Small Lung Cancer
Brief Title: Pulmonary Rehabılıtatıon Wıth Non-Small Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Kardelen HATIMOĞULLARI, physiotherapist, Hasan Kalyoncu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018/09
Record Dates: First submitted 2022-02-25; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Lung Cancer; Lung Cancer, Small Cell
Keywords: Lung Cancer; Pulmonary Rehabilitation; Aerobic Exercise; Physiotherapy and Rehabilitation; Oncological Rehabilitation
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: Single group 30 individuals were included in the study. Surgery, adjuvant chemotherapy and radiotherapy processes of all patients included in the study were completed. Patients between the ages of 18-65 and in remission period were included in the study. Patients with suspected pregnancy, diabetes mellitus, metastatic patients, and patients with acute and chronic infections were excluded from the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary Rehabilitation (Experimental): Pulmonary rehabilitation program will be applied 3 days a week at 40-60% of submaximal heart rate for a total of 8 weeks. Diaphragmatic breathing, pursed lips and segmental breathing exercises will be applied to the patients in the presence of a physiotherapist. Walking and aerobic exercise training will be given.
  Interventions: Other: Pulmonary Rehabilitation

INTERVENTIONS:
Other: Pulmonary Rehabilitation — 1-Pulmonary Rehabilitation: Pulmonary rehabilitation program was applied at 40-60% of submaximal heart rate, 3 days a week for a total of 8 weeks. Diaphragmatic breathing, pursed lip breathing and segmental breathing exercises were practiced with the patients in the company of a physiotherapist. Walking and aerobic exercise training was given.

SUMMARY:
The aim of our study is to investigate the effects of pulmonary rehabilitation on respiratory tests and quality of life in patients with early and locally advanced NSCLC who received chemotherapy regardless of whether the investigators had undergone surgical treatment.

DETAILED DESCRIPTION:
Patients with lung cancer often have concomitant lung and heart comorbidities that limit their cancer treatment options. For example, in the last prevalence study that included patients with newly diagnosed lung cancer, 73% of whom were men and 53% were women, there was clinically significant COPD. This patient population has shortness of breath, decreased physical capacity, low muscle condiction, and poor exercise tolerance.

Pulmonary rehabilitation is an intervention that has a scientific basis and is used systematically, aiming to optimize individual daily functions and health-related quality of life in patients with morbidity due to chronic diseases measured by clinical or physiological methods.

The effectiveness of pulmonary rehabilitation is well known in the treatment of patients with COPD and in the perioperative lung transplant preparation period. Studies lead to a significant increase in preoperative pulmonary rehabilitation exercise capacity, dyspnea and health-related quality of life.

The aim of our study is to investigate the effects of pulmonary rehabilitation on respiratory tests and quality of life in patients with early and locally advanced NSCLC who received chemotherapy regardless of whether the investigators had undergone surgical treatment.

This study was conducted with outpatients who were diagnosed with small cell lung cancer between 2021-2022, who were approved by the oncologist and physical therapist to participate in a physiotherapy and rehabilitation program. Permission for the study was obtained from the Non-Interventional Local Ethics Committee (decision dated 20.11.2018 and numbered 2018/34). The study was conducted in accordance with the Helsinki Declaration of Patient Rights. Individuals were informed about the study and a written informed consent form was signed by the individuals who volunteered to participate.

Participants Thirty patients aged 18-65 years in remission were included in the study. Surgery, adjuvant chemotherapy and radiotherapy processes of all patients included in the study were completed. Patients with suspected pregnancy, diagnosis of diabetes mellitus, patients in metastatic period, and patients with acute/chronic infection were excluded from the study.

Evaluation The patients' age, gender, height and body weight, medical history and family history information, education status, income level, smoking (pack/year), place of residence, admission to the emergency department in the last year, number of hospital admissions and hospitalizations, and medication used The information was recorded from the patients and their files. Participation of individuals in regular physical activity was questioned. In addition, pre- and post-treatment pain was evaluated using the visual analog scale (VAS).

The evaluations applied to the patients in our study;

1. Posture Analysis
2. Normal Joint Movement and Evaluation of Muscle Shortness
3. Muscle Test
4. Six Minute Walking Test
5. Physical Activity Level
6. Dyspnea Severity
7. Quality of Life
8. Fatigue Evaluation

Applied Treatments;

1. Respiratory Exercises
2. Walking Training
3. Aerobic exercise training

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-65, must be in remission.
* Surgery, adjuvant chemotherapy and radiotherapy processes must be completed.

Exclusion Criteria:

* Those with suspected pregnancy
* Diabetes mellitus diagnosis
* Patients in the metastatic period
* Patients with a diagnosis of acute/chronic infection were excluded from the study.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2022-05-02 (Estimated); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-09-02 (Estimated)

PRIMARY OUTCOMES:
Chance from baseline in posture analysis score | 8 week
  Posture score is going to be assess by posture analysis form to determine change from baseline.

SECONDARY OUTCOMES:
Physical Activity Level | 8 week
  Physical Activity is going to be assess by Physical Activity Questionnaire to determine change from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu Univercity, Gaziantep, Turkey (Türkiye)